CLINICAL TRIAL: NCT04158414
Title: Applying PET/MR in Oncology - a Prospective Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-19-ES-0568-CTIL
Record Dates: First submitted 2019-10-29; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Lymphoma; Nasopharyngeal Cancer; Esophageal Cancer; Cervical Cancer; Hepatobiliary Cancer; Pancreatic Cancer; Sarcoma; Prostate Cancer
MeSH Terms: conditions — Lymphoma; Nasopharyngeal Neoplasms; Esophageal Neoplasms; Uterine Cervical Neoplasms; Pancreatic Neoplasms; Sarcoma; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Different types of cancer Patients (Experimental): Lymphoma,Nasopharyngeal Cancer; Esophageal Cancer, Cervical cancer; Hepatobiliary and pancreatic cancer; Sarcoma; Prostate Cancer
  Interventions: Diagnostic Test: PET/MR scan

INTERVENTIONS:
Diagnostic Test: PET/MR scan — 500 cancer patients referred to PET-CT assessment will undergo PET/MR scan as well, and the net data will be compared. The overall data will be investigated in groups and subgroups of patients that share similar clinical characteristics and represent cancer patients in different time points during the natural history of their disease. Data analysis will be performed both visually and quantitatively using different MR and PET parameters according to the patient group. Specific populations will be detailed in the next sections per malignancy.

SUMMARY:
Cancer is a global health issue. According to the World Health Organization, Cancer is the second leading cause of death globally, and is responsible for an estimated 9.6 million deaths in 2018. In Israel, more than 30,000 new cases of cancer were diagnosed, and more than 11,000 deaths were cancer-related during 2016.

Imaging plays a pivotal role in cancer management, and multiple techniques are used in all phases of cancer management. The overall morphological, structural, metabolic and functional information obtained in imaging is used for improved individualized therapy planning. Different imaging modalities are available during different time points in the natural history of different malignancies:

Early detection of cancer through screening based on imaging is probably a major contributor to a reduction in mortality for certain cancers .

Once a diagnosis is made, determining the clinical stage of cancer, meaning the extent of the disease before any treatment is given, is a critical element in determining appropriate treatment based on the experience and outcomes of groups of previous patients with similar stage . Precise clinical staging of cancer is crucial. Not only that this clear non-ambiguous description is a key factor that defines prognosis, it is also a chief component of inclusion, exclusion, and stratification criteria for clinical trials. Several cancer staging systems are used worldwide. The most clinically useful staging system is the tumor, node, and metastasis (TNM) staging system developed by the American Joint Committee on Cancer (AJCC) in collaboration with the Union for International Cancer Control (UICC). The AJCC TNM system classifies cancers by the size and extent of the primary tumor (T), involvement of regional lymph nodes (N), and the presence or absence of distant metastases (M). There is a TNM staging algorithm for cancers of virtually every anatomic site and histology, with the primary exception of pediatric cancers. The clinical TNM (cTNM) classification should be used to determine correctly the clinical stage of cancer and to help guide primary therapy planning.

DETAILED DESCRIPTION:
Stage may be defined at several time points during the monitoring period of cancer patients. When using imaging obtained during the relevant time frame, one may use one of the other TNM categories to stage correctly the cancer:

For example, imaging is of high value in assessing therapy response during and after systemic and/or radiation therapy is given . Using imaging data and the clinical posttherapy TNM classification (ycTNM) is helpful in determining the patient's response to treatment.

In case a patient is given the systemic therapy as a neoadjuvant therapy before a planned curative surgery, imaging may categorize the patient as a responder vs non-responder. If categorized as an early non-responder, another therapy or an upfront surgery may be advised, while eliminating therapy toxicity. If imaging, however, supports major response to treatment, more conservative treatment and avoidance of surgical intervention may be considered and change patients quality of life dramatically.

In patients given a systemic therapy as a curative or a palliative therapy, assessing the response via imaging is crucial as well - if imaging studies support a progressive disease, changing therapy protocol is advised. In a disease controlled by the therapy, imaging may aid in guiding follow-up schedule, lifestyle and medical management.

In the context of therapy response assessment, imaging is also important in assessing side effects of the therapy. Imaging may identify radiation-induced injuries, and may recognize pathologies associated with chemotherapy, biologic and immunotherapy.

Imaging is also critical when recurrence of malignant disease is suspected. In such cases, when signs or symptoms suggest local recurrence, or when raised level of a tumor marker is documented, different imaging techniques can dramatically guide restaging of the disease using the recurrence-TNM classification (rTNM). In such cases imaging may localize the recurrent disease and may guide surgical/radiation/systemic therapy .

Different imaging modalities allow assessment of virtually every cancer site and in every time frame during the continuum of the disease. Imaging aids in assessing tumor's size, location, and relationship to normal anatomic structures, as well as the existence of nodal and/or distant metastatic disease. Among the most commonly used imaging modalities are computed tomography (CT), magnetic resonance (MR) imaging, positron emission tomography (PET) and ultrasound. In addition to providing key information for assigning the T, N, and M categories, imaging is invaluable for guiding biopsies and surgical resections.

PET imaging has revolutionized the imaging evaluation of cancer . By exploiting biochemical and physiologic differences between tumor cells and normal tissues , PET imaging has become

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed in One of the cancers being investigated.
2. Only in Sarcoma:20 children and adults with newly diagnosed sarcomas. Children will be included if can perform the study without sedation, and with written parental approval.

Exclusion Criteria:

1. Patients younger than 18 years.
2. Pregnancy/
3. Patients contraindication to MRI or to intravenous gadolinium injection.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-11-28 (Estimated); Primary Completion 2020-01-28 (Estimated); Study Completion 2021-11-28 (Estimated)

PRIMARY OUTCOMES:
Patients who preformed PET/MR and PET/CT in clinical staging and monitoring of different cancer types will be measured and reported number of Participants in staging and different between their scans/ | 1 year

IPD SHARING:
Plan to Share IPD: Undecided